CLINICAL TRIAL: NCT03954353
Title: Effect of Cholesterol Level on Postoperative Acute Kidney Injury of Non-cardiac Surgeries
Status: Completed | Type: Observational
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Yan Zhou, MD, Principal Investigator, Peking University First Hospital
Other Study IDs: ECAKI
Record Dates: First submitted 2019-05-16; First posted 2019-05-17 (Actual); Last update posted 2019-07-09 (Actual); Status verified 2019-07

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Preoperative serum cholesterol level may influence occurrence of postoperative acute kidney injury of cardiac surgeries. However, the effect of Preoperative serum cholesterol level for non cardiac surgery remains unknown. This study aimed to explore the effect in non-cardiac surgical population.

ELIGIBILITY:
Inclusion Criteria:

adults elective non-cardiac surgery

Exclusion Criteria:

cardiac surgeries kidney surgeries obstetric surgeries local infiltration anesthesia perioperative data missing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adults (age ≥ 18 years old) who underwent elective non-cardiac surgery from January 1, 2012, to December 31, 2017.
Sampling Method: Non-Probability Sample
Enrollment: 78888 (Actual)
Dates: Start 2019-05-17 (Actual); Primary Completion 2019-06-05 (Actual); Study Completion 2019-06-06 (Actual)

PRIMARY OUTCOMES:
post-operative acute kidney injury within 30 days in the hospital | 30 days postoperatively in hospital
  It was defined by patient's postoperative serum creatine increase no less than 26.5 μmol/l within 48 hours, or 1.5 times from baseline within the 7 days after surgery or initializing blood dialysis.

CONTACTS AND LOCATIONS:
Locations (1):
- First hospital Peking University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zhou Y, Yang HY, Zhang HL, Zhu XJ. High-density lipoprotein cholesterol concentration and acute kidney injury after noncardiac surgery. BMC Nephrol. 2020 Apr 25;21(1):149. doi: 10.1186/s12882-020-01808-7. PMID 32334566